



# Public Benefit and Privacy Panel for Health and Social Care

## **Application Form**

| Application Control | | | |
|---|---|---|---|
| Applicants should not fill out this | Applicants should not fill out this section | | |
| Application Coordinator | Dionysis Vragkos | | |
| Application Number | 1516-0370 | Submitted Date | 07/09/2016 |
| Applicant Name | Richard Peter Gerardus ten Broek | | |
| Proposal Name | Adhesion-related hospital readmissions after abdominal and | | |
| | pelvic surgery: An update of the SCAR studies | | |





#### Contents

| Note to Applicants | 2 |
|---|---|
| Section 1 – People | 3 |
| Section 2 – Organisations & Bodies | 7 |
| Section 3 – Overview | 10 |
| Section 4 – Data & Data Subjects | 18 |
| Section 5 – Methodology & Data Processing | 23 |
| Section 6 – Declaration | 29 |
| Section 7 - Supporting Evidence | 30 |
| Appendix A – Reference lists for applicants | 31 |
| Appendix B –The Caldicott Principles & the Data Protection Principles (& Schedules) | 33 |

### **Note to Applicants**

### Prior to completing your application form you should:

- Contact the eDRIS Team, who will assist you <u>Nss.edris@nhs.net</u> or by phone on 0131 275 7333
- Read and understand the separate Guidance for Applicants

Your application should be typed, not handwritten. Your eDRIS application coordinator will inform you how to submit your application form and any supporting evidence. Before submitting your completed application, you should ensure that:

- All relevant sections of the application are complete
- Relevant supporting evidence is attached
- Individuals named on the form have read and approved its submission

<u>Please note</u> that submitted applications may be circulated to panel members, administrative colleagues, NHSScotland information governance and information security colleagues, Caldicott Guardians, the CHI Advisory Group and, where appropriate, non-NHS Scotland colleagues from a variety of participating partner bodies, in the course of processing. You must make your eDRIS application coordinator aware of any confidential or sensitive information contained in your application which you would consider inappropriate for circulation in such a manner. Your application could be subject to disclosure or partial disclosure under the Freedom of Information (Scotland) Act, and will be retained in line with NHSScotland information policy.





## Section 1 - People

| 1.1 | Applicant Please read section 1.1 of the guidance | |
|---|---|---|
| 1.1.01 | Full Name: | Richard Peter Gerardus ten Broek |
| 1.1.02 | Title: | MD, PhD |
| 1.1.03 | Position: | Post-doctoral researcher, Project coordinator |
| 1.1.04 | Professional Registration No. | If applicable |
| 1.1.05 | Organisation Name: | Radboud University Medical Center, Nijmegen, the |
| | | Netherlands - department of Surgery |
| 1.1.06 | Address: | PO box 9101 |
| 1.1.07 | Postcode: | 6500 HB, Nijmegen, the Netherlands |
| 1.1.08 | Telephone Number: | +31636304310 |
| 1.1.09 | Email: | Richard.tenBroek@radboudumc.nl |
| 1.1.10 | Do you have an NHS | No |
| | contract/honorary contract? | |
| 1.1.11 | Provide details of the most re- | details of the most recent information governance training undertaken - a list of |
| | training courses is included at | Appendix A, and you should particularly indicate if you |
| | have undertaken any of those | listed |
| | Name of course: | MRC Research Data and Confidentiality online module |
| | Link to course content: | MRC Research Data and Confidentiality online module |
| | Institution: | Medical research Council |
| | Date completed: | May 12 2016 |

| 1.2 | Clinical Sponsor/Lead Please read section 1.2 of the guidance | |
|---|---|---|
| 1.2.01 | Full Name: | Ewen A Griffiths MD, FRCS |
| 1.2.02 | Title: | Consultant Upper GI and General Surgeon, |
| 1.2.03 | Position: | Clinical sponsor |
| 1.2.04 | Professional Registration No.: | GMC 4732039 |
| 1.2.05 | Organisation Name: | Queen Elizabeth Hospital, Birmingham |
| 1.2.06 | Address: | University Hospitals NHS Foundation Trust |
| | | Edgbaston, Birmingham, UK |
| 1.2.07 | Postcode: | B15 2TH |
| 1.2.08 | Telephone Number: | 0121 3715883 |





| 1.2.09 | Email: | Ewen.griffiths@uhb.nhs.uk |
|---|---|---|
| 1.2.10 | Does this person have an NH | S Yes |
| | contract/honorary contract? | |
| 1.2.11 | Provide details of the most re | cent information governance training undertaken - a list of |
| | training courses is included at | t <u>Appendix A</u> , and you should particularly indicate if this |
| | person has undertaken any o | f those listed |
| | Name of course: | MRC Research Data and Confidentiality online module |
| | Link to course content: | MRC Research Data and Confidentiality online module |
| | Institution: | Medical research Council |
| | Date completed: | 1 <sup>st</sup> Aug 2016 |

| 1.3 | Information/Data Custodian F | Information/Data Custodian Please read section 1.3 of the guidance |
|---|---|---|
| 1.3.01 | Full Name: | Same as applicant |
| 1.3.02 | Title: | |
| 1.3.03 | Position: | |
| 1.3.04 | Professional Registration No.: | If applicable |
| 1.3.05 | Organisation Name: | |
| 1.3.06 | Address: | |
| 1.3.07 | Postcode: | |
| 1.3.08 | Telephone Number: | |
| 1.3.09 | Email: | |
| 1.3.10 | Does this person have an NHS | Choose an item. |
| | contract/honorary contract? | |
| 1.3.11 | Provide details of the most recent information governance training undertaken - a list of | |
| | training courses is included at A | Appendix A, and you should particularly indicate if this |
| | person has undertaken any of those listed | |
| | Name of course: | |
| | Link to course content: If | applicable |
| | Institution: | |
| | Date completed: | |

# **1.4 Others with access to identifiable or potentially identifiable data** *Please read section 1.4* of the guidance





| Complete this section if applicable – for each additional person | | | | | | |
|---|---|---|---|---|---|---|
| Full Name: | Pepijn Krieler | 1 | Telephone or | Email: | +3161321 | 18398 |
| Organisation: | Radboud Univ | versity Medical | Position: | | PhD Stud | ent |
| | Center | | | | | |
| Professional | Z478129 | | NHS contract | / | No | |
| Registration No: | | | honorary cont | tract? | | |
| IG Training - Name of course: MRC Researc | | MRC Research | Data and Con | nfidentia | lity online n | nodule |
| IG Training - Link to course: MRC Research | | ch Data and Confidentiality online module | | <u>nodule</u> | | |
| IG Training - Institution: | | Medical resear | rch Council Date completed: 8 <sup>th</sup> AUC | | 8 <sup>th</sup> AUG 2017 | |

| Full Name: | Janienke van | Lier | Telephone or | Email: | +3161321 | 18398 |
|---|---|---|---|---|---|---|
| Organisation: | Radboud University Medical | | Position: | | PhD Stud | ent |
| | Center | | | | | |
| Professional | Z516230 | | NHS contract | / | No | |
| Registration No: | | | honorary cont | tract? | | |
| IG Training - Name of course: MRC Research | | Data and Con | ıfidentia | lity online n | nodule | |
| IG Training - Link to course: MRC Research | | h Data and Confidentiality online module | | nodule | | |
| IG Training - Institution: Medi | | Medical resear | ch Council | Date c | ompleted: | |

| 1.5 Others Please read section 1.5 of the guidance | | | |
|---|---|---|---|
| Complete this | Complete this section if applicable – for each additional person | | |
| Full Name: | Michael Parker | Involvement in | Principal investigator, Study |
| | | Proposal: | design |
| Organisation: | Royal College of Surgeons | Position: | Emeritus Professor in Surgery, |
| | | | study steering group |

| Complete this section if applicable – for each additional person | | | |
|---|---|---|---|
| Full Name: | Harold Ellis | Involvement in | Study design |
| | | | , , |
| | | Proposal: | |
| Organisation: | Kings college London | Position: | Emeritus professor, study |
| - 5 | 3 | | · |
| | | | steering group |
| Complete this section if applicable – for each additional person | | | |
| complete the ecotion if applicable for each additional percent | | | |





| Full Name: | Harold Ellis | Involvement in | Study design |
|---|---|---|---|
| | | Proposal: | |
| Organisation: | Kings college London | Position: | Emeritus professor, study |
| | | | steering group |





## Section 2 – Organisations & Bodies

| 2.1 | Organisation or Body Leading Proposal Please read s | section 2.1 of the guidance |
|---|---|---|
| 2.1.01 | Organisation or Body Name: | If the organisation here is an |
| | Dutch Adhesion Group | NHSScotland board, note this |
| | (Research workgroup linked to the Dutch college of | and go directly to question |
| | gastro-intestinal surgeons and Dutch college of | 2.1.4 |
| | gynaecologists and obstetricians) | |
| 2.1.02 | Is this organisation or body a registered data | No |
| | controller? If 'Yes', provide Data Protection Registration | |
| | Number: | |
| 2.1.03 | Is this a commercial organisation or body? | No |
| 2.1.03a | If 'Yes', please provide a full explanation of the | If applicable |
| | organisation or body's activity and industry sector, | |
| | including any previous experience of using | |
| | NHSScotland data - append supporting documentation | |
| | as appropriate | |
| 2.1.04 | Is this organisation or body wholly funding or paying for | Yes |
| | the costs of conducting the proposal? | |

| 2.2 | Organisation or Body Funding Proposal Please read section 2.2 of the guidance | |
|---|---|---|
| Complete the following section if you answered 'No' to question 2.1.4 | | |
| 2.2.01 | Organisation or Body Name: | If the organisation here is an |
| | | NHSScotland board note this |
| | | and, go directly to section 2.3 |
| 2.2.02 | Is this organisation or body a registered data | No |
| | controller? If 'Yes', provide Data Protection Registration | |
| | Number: | |
| 2.2.03 | Is this organisation or body a commercial organisation? | No |
| 2.2.03a | If 'Yes', please provide a full explanation of the | |
| | organisation or body's activity and industry sector, | |
| | including any previous experience of using | |





| NHSScotland data - append supporting documentation |
|----------------------------------------------------|
| as appropriate |





| 2.3 Other Relevant Organisations or Bodies Please read section 2.3 of the guidance | | |
|---|---|---|
| Complete this section if applicable | | |
| Organisation Name | Nature of Business/Sector | Nature of interest in proposal |
| Radboud University Medical | University Medical Center | University supporting proposal |
| Center, Nijmegen, the | | and facilitating the applicant |
| Netherlands | | |





## Section 3 – Overview

| 3.1 | Proposal Essentials Please read section 3.1 of the guidance | | |
|---|---|---|---|
| 3.1.01 | Proposal title/name: | | Adhesion-related hospital |
| | | | readmissions after abdominal and |
| | | | pelvic surgery: An update of the |
| | | | SCAR studies |
| 3.1.02 | Is this proposal an extension or renewal or | f an | No |
| | existing approval (for example to conduct | a study | |
| | over a wider geographic area or for a long | er | |
| | period of time)? Please provide details, inc | clude | |
| | the reference number of the original appro | val, | |
| | and summarise the changes requested | | |
| 3.1.03 | Is this new proposal related to a previous | | No |
| | application (approved or not)? Please give | ) | |
| | details, indicate if this is a resubmission, in | ncluding | |
| | the reference number of the original subm | ission | |
| 3.1.04 | What is(are) the substantive purpose(s) of | the prop | osal? (tick all that apply) |
| | □ Patient Care □ | Resear | rch |
| | □ Audit □ | Perforn | nance Monitoring/Management |
| | ☐ Service Planning/Improvement ☐ | Health/ | Social Care Administration |
| | ☐ Systems Implementation/Testing ☐ | Training | g/Education |
| | ☐ Quality (Clinical, Educational, etc) | | |
| | If other clearly defined purpose, please give | e details | • |
| 3.1.05 | Does the proposal require the use of inform | mation | No |
| | which can identify or potentially identify | | |
| | individuals? | | |
| 3.1.06 | Access is being requested to data from wh | nich sourc | ces? (tick as many as are relevant) |





| | □ A single NHS Scotland Board (excluding NSS) |
|---|---|
| | □ NHS National Services Scotland |
| | ☐ More than one NHS Scotland Board |
| | ☐ More than one NHS Scotland system/database |
| | ☐ Community Health Index (CHI) database |
| | □ NHS Central Registry |
| | If other, please give details: |
| 3.1.07 | Provide a full, clear concise outline of the proposal background – describe why it is |
| | needed, aims and objectives and envisaged benefits to the public and/or patients: |
| | Adhesion formation is the most common cause for long – term complications in |
| | abdominal surgery. Abdominal surgery is performed by a multitude of specialist, |
| | including general surgeons, gynaecologists, vascular surgeons and urologists. In |
| | Scotland, like many other developed countries, adhesion- related complications cause a |
| | huge burden of morbidity. Adhesion-related complications comprise various clinical |
| | entities such as small bowel obstruction, chronic pain and female infertility. |
| | In 1999 Prof. Ellis demonstrated in the SCAR studies, using data from the Scottish |
| | National Health Service record linkage database, that as many as 34.6% of patients |
| | undergoing abdominal surgery are readmitted for complications directly or possibly |
| | related to adhesion formation in 10 years after surgery. |
| | Since this landmark study a number of strategies were introduced to reduce adhesion |
| | formation. First are the so-called 'anti-adhesion' barriers. Almost simultaneously there |
| | has been the rise of minimal invasive surgery. Minimal invasive surgery is associated |
| | with less extensive peritoneal injury and adhesion formation. |
| | While minimal invasive surgery became adopted quickly, the use of anti-adhesion |
| | barriers remains marginal. Many surgeons therefore feel that with laparoscopy further |
| | adhesion prevention is not necessary, despite some evidence that incidence of |
| | adhesion- related complications is still considerable. |





To evaluate the impact of laparoscopic surgery on adhesion- related formation, we are planning to perform an update of the SCAR studies to recent years in which a large number of laparoscopic surgeries have been performed. Comparison of readmissions for adhesion- related complications after open and laparoscopic surgery will be made. The study will provide an estimate of the current burden of adhesion-related morbidity in Scotland, which could also serve as a model for the current burden in other European countries. Further such estimate can be used to model the impact of further implementation of anti-adhesion barriers on adhesion-related morbidity and healthcare costs in both Scotland and abroad.

3.1.08 Provide a full, clear and concise outline of the proposal design, listing: data sources; sample size; inclusion/exclusion criteria (eg involvement in trial/survey; health event, etc); relevant date range; need for identifiable or potentially identifiable data; requirement for a matched control cohort etc.

We intend to use the Scottish National Health Service record linkage capabilities. Inclusion criteria are all patients undergoing initial abdominal or pelvic surgery between June 2009 and June 2011. Selection will be made by OPCS-4 codes related to the admission. A list of relevant codes can be found in the appendix. We choose for these years to allow inclusion of an incident population in a time that laparoscopic surgery had already been implemented and that allows for 4 to 5-years of follow-up.

We will exclude patient who had had abdominal or pelvic operation in the 5 years before 2009, as pre-existing adhesions from this prior surgery might influence results. There are no further exclusion criteria.

For analyses patients will be grossly divided in three groups of anatomical location of the surgery: hindgut, female reproductive tract, and foregut or other. Within each group subgroups of laparoscopic and open procedures will be made.

We expect approximately 70,000- 100,000 patients to have had abdominal or pelvic surgery in the period June 2009- June 2011. Approximately 25,000 are expected to have had prior abdominal surgery in the previous 5 years. Thus, we expect an incident population of 45,000 to 75,000 to be included in the study.





For the study we will analyse re-admission in the years following surgery that are directly related to adhesions, possibly related to adhesions, and readmission with surgery that might be complicated by adhesions. For this purpose we will need a patient identifier that allows to link readmissions to the initial surgery. The data can be anonymized so that the identifier represent just a random number. As baseline characteristics we will only require age and sex. No further potentially identifiable data such as birth date, postal code or NHS number is required. From the initial admission with abdominal or pelvic surgery we need ICD- 10 codes and OPCS- 4 codes describing the type of surgery performed as well as information whether the operation was performed laparoscopic ally or open. This same set of information is needed for any readmission in follow-up. Further we need the time interval (in months) between the index operation and the readmission. Only readmissions coded by one or more relevant ICD-10 or OPCS-4 code need to be included. For a readmission to be classified as directly related to adhesions, an explicit adhesion reference was required in the operative OPCS-4 or diagnostic ICD-10 coding. Adhesions might however not always be coded, especially not if readmission goes without surgery. For example, a conservative treated small bowel obstruction might only be coded as abdominal pain, nausea, and vomiting. Therefore we will define a broader set of operative codes and diagnostic codes that might indicate a possibly adhesion-related complication. Data from follow-up is requested to the latest date from which a complete record can be extracted.

3.1.09 Does the proposal have implications for, or target, sensitive groups or vulnerable populations? Please give details

No

3.1.10 Does the proposal seek to use information exclusively about deceased persons? Please give details

No





| 3.1.11 | Have any members of the public/lay representatives been involved in the proposal |
|---|---|
| | design? Please give details |
| | No |
| 3.1.12 | Has any peer review of the proposal been undertaken? Please give details (for example |
| | formal review by a peer organisation or funding body, informal internal review, review by |
| | a third party) |
| | Informal internal review has been performed within the Radboud University Medical |
| | Center, department of Surgery. The research proposal and internal funding for |
| | performing the study were approved. |
| 3.1.13 | Is there any commercial aspect or dimension to the proposal or its outcomes? Please |
| | give details |
| | No |

| 3.2 | 3.2 Proposal Geography Please read section 3.2 of the guidance |
|---|---|
| | Local/Regional (relating to one or more specific areas within Scotland) |
| $\boxtimes$ | National (relating to the whole of Scotland) |
| | UK-wide (relating to the whole of the UK, or to UK regions outside Scotland) |
| | International (relating to areas within the EEA) |
| | International (relating to areas beyond the EEA) |

## 3.3 Proposal Duration and Frequency Please read section 3.3 of the guidance





| 3.3.01 | What is the proposed duration of the proposal? | We now requested for access to the |
|---|---|---|
| | | data until 2019-12-31, for the purpose |
| | | of answering a few questions of the |
| | | editorial team of Lancet on the |
| | | presentation of the data (e.g. adding |
| | | standard deviations to data |
| | | presented) |
| 3.3.02 | Does the proposal require updates of | no |
| | information at regular intervals? Please give | |
| | details | |
| 3.3.03 | Are you seeking approval to iterate the proposal | no |
| | (ie the whole project, audit or study) at regular | |
| | intervals? Please give details | |

| 3.4 | Statutory and Regulatory Context Please read section 3.4 of the guidance | |
|---|---|---|
| 3.4.01 | Does your proposal have a statutory or | NO |
| | regulatory justification - is the proposal | |
| | responding to a statutory or regulatory | |
| | instruction, duty or order? Please give details | |
| 3.4.02 | Which Data Protection Act schedule 2 and | Schedule 2: |
| | schedule 3 conditions are relevant? (a list of | Condition 3; the use of patient |
| | conditions can be found at Appendix B) | identifying data is not necessary to |
| | | carry out the research. The linking |
| | | code can be anonymized using a |
| | | random number. The researcher |
| | | therefore do not need identifying data |
| | | for carrying our analyses. Also the |
| | | use of data which is not directly |
| | | identifiable is minimized, by |
| | | requesting a minimum in baseline |
| | | characteristics and only data from |
| | | readmissions with a relevant code. |
| | | Schedule 3, Condition 8: |





| | | The processing is necessary for |
|---|---|---|
| | | medical researcher, and analyses is |
| | | undertaking by health professional |
| | | who completed information |
| | | governance training. |
| 3.4.03 | Are there any relevant information sharing | No |
| | agreements, protocols or contracts in place | |
| | which support your proposal? Please give | |
| | details and attach as supporting documentation | |
| | if available | |
| 3.4.04 | Has a Privacy Impact Assessment been carried | Yes, see attachment. Privacy risk can |
| | out which supports your proposal? Please give | be adequately eliminated. |
| | details and attach as supporting documentation | |
| | if available | |
| 3.4.05 | Has local Caldicott approval been given for your | No |
| | proposal at a local level? Please give details | |
| 3.4.06 | Are approvals from Caldicott Guardians outside | No |
| | Scotland pending or received? Please give | |
| | details | |

| 3.5 | Research and Ethics Governance Please read section 3.5 of the guidance | |
|---|---|---|
| 3.5.01 | Has your proposal sought research/ethics | Yes |
| | approval? | |
| 3.5.01a | If yes, please provide committee details and | Radboud University medical Center- |
| | status of approval (ie pending, approved, etc). | Institutional review board |
| | Please attach as supporting documentation if | PO box 9101 |
| | available | 6500 HB, Nijmegen, the Netherlands |
| | | T +3124 361 31 54 |
| | | E:commissiemensgebondenonderzoek@ |
| | | RadboudUMC.nl |
| | | - approved - |
| 3.5.01b | If no, please explain why research/ethics | |
| | approval is not sought: | |





| 3.6 | Safe Havens Please read section 3.6 of the guida | nce |
|---|---|---|
| 3.6.01 | Do you intend to access the data requested | Yes, |
| | exclusively through a safe haven listed at | NHS NSS ISD Electronic Data |
| | Appendix A? Please provide details of which safe | Research Innovation Service (@Farr |
| | haven/s | <u>Institute</u> ) |
| 3.6.02 | If you applying to use NHS NSS data and you do | Not applicable |
| | not intend to do this through the National Safe | |
| | Haven, please explain why | |





## Section 4 – Data & Data Subjects

| 4.1 Data yet to be collected Please read section 4.1 of the guidance | | |
|---|---|---|
| Not applicable | | |
| Dataset/source<br>Name | Collection by (whom)? | Explicit consent sought? If Yes, describe how explicit consent being sought – provide copies of |
| | | participant consent/registration forms, etc. If No, explain why consent is not being sought (eg |
| | | impractical, risk associated with seeking consent, etc) |

| 4.2 All Other Datase | 4.2 All Other Datasets / sources Please read section 4.2 of the guidance | |
|---|---|---|
| Dataset/source | Data Controller (Organisation) Original purpose compatible with | |
| Name | | proposal? |
| Scottish Morbidity | National Services Scotland | Yes |
| Record (SMR01) | | |
| NRS Deaths | NRS | Yes |
| CHI Database | NHS Boards | Yes |

How were individuals originally informed of the use of their data? (if known)

Project specific consent was impractical for this study because of large size of the survey group and patients are not contacted. However:

- a) no identifiable patient data will be disclosed
- b) the necessary linkage will be performed by data controllers from the NHS Scotland board, that already hold the data. After linkage the data will be anonymised.
- c) the medical research serves public interest as outlined under 3.1.07.

The final dataset for analysis will not hold data that could result in indirect identification.

For existing dataset/sources for which the data controller is not an NHSScotland board, please append evidence of the data controllers permission to use the data

## **4.3 Data Variables** Please read section 4.3 of the guidance





| Dataset/source | Variable | Time Period/Range | Processing only? |
|---|---|---|---|
| Name | | | |
| Anonymised ID | | | |
| Scottish Morbidity | CHI | 2004- Dec 2016 | Yes |
| Record (SMR 01) | | | |
| Scottish Morbidity | Date of admission | 2004- Dec 2016 | No |
| Record (SMR 01) | | | |
| Scottish Morbidity | Sex | 2009- Dec 2016 | No |
| Record (SMR 01) | | | |
| Scottish Morbidity | Age (Date of admission- | 2009- Dec 2016 | No |
| Record (SMR 01) | birth date) | | |
| Scottish Morbidity | ICD-10 codes | 2009- Dec 2016 | No |
| Record (SMR 01) | | | |
| Scottish Morbidity | OPCS-4 codes | 2009- Dec 2016 | No |
| Record (SMR 01) | | | |
| Scottish Morbidity | Duration since index | 2009- Dec 2016 | No |
| Record (SMR 01) | operation (date of | | |
| | admission from | | |
| | readmission - date of | | |
| | admission from index | | |
| | operation) | | |
| Scottish Morbidity | Details of operation - | 2009- Dec 2016 | No |
| Record (SMR 01) | laparoscopic/ open | | |
| Scottish Morbidity | End of follow-up (month) | 2004- Dec 2016 | No |
| Record (SMR 01) | (Date of end of follow-up, | | |
| | typically June 2016; | | |
| | however some patient | | |
| | might not complete follow- | | |
| | up because of mortality or | | |
| | migration) | | |
| Scottish Morbidity | Continuous Inpatient Stay | 2009- Dec 2016 | No |
| Record (SMR 01) | | | |
| CHI Database | Migration Month / year | 2004- Dec 2016 | No |





| NRS Deaths | Patient alive or death by | 2004- Dec 2016 | No |
|---|---|---|---|
| | end of follow-up | (measured in | |
| | | months, no date | |
| | | provided) | |
| Please justify your nee | d for identifiable or potential | ly identifiable variables | : |
| Identifiable data is only needed during the processing of data. Data will be collected during a range | | | |
| of 5 years from index s | of 5 years from index surgery. Patients with a relevant OPCS-4 code as listed in the appendix are | | |
| selected, if no prior su | ich operation was found in | the five years previous | to the index operation. |
| Identifiable information | n, NHS number and birth | date are needed duri | ng processing to select |
| reoperations that are of | definitely or potentially relate | ed to adhesion in patie | ents following their index |
| surgery. After processing these data can be removed. Age is potential risk factor for adhesions and | | | |
| will therefore be calculated. | | | |

| 4.4 | NRS/NHSCR Data Sources Please read section 4.4 of the guidance | | |
|---|---|---|---|
| Complet | e this section if access to NHSCR is requir | ed, or if there is any | National Records of |
| Scotland | l involvement | | |
| 4.4.01 | Does the proposal require access to NHS | Central Registry | No |
| | as a sampling frame for cohorts? | | |
| 4.4.02 | Does the proposal involve flagging of indi- | viduals on the | Choose an item. |
| | NHSCR for long term follow up? | | |
| 4.4.03 | If yes, is flagging necessary: | | |
| | ☐ To trace and contact individuals throughout the UK? | | |
| | ☐ To be informed of fact and cause of death? | | |
| | ☐ To be informed of the incidence of on-going cancers? | | |
| | ☐ To be informed of emigrations prospectively and retrospectively? | | |
| 4.4.04 | Is any other NRS involvement required? | | |
| | Please provide details | | |

| 4.5 | Making Contact with Individuals Please read section 4.5 of the guidance | |
|---|---|---|
| 4.5.01 | Is any direct contact with any group of individuals required? If No | |
| | Yes, please provide details below | |
| | Contact Group and Method of contact | Contact by (whom) |





| | ☐ Hospital Consultants | □ Letter | ☐ Phone | ☐ Other | |
|---|---|---|---|---|---|
| | | | | (specify): | |
| | ☐ Other NHSS Staff | □ Letter | ☐ Phone | □ Other | |
| | | | | (specify): | |
| | ☐ General Practitioners | □ Letter | ☐ Phone | □ Other | |
| | | | | (specify): | |
| | □ Patients/Public | □ Letter | ☐ Phone | □ Other | |
| | | | | (specify): | |
| | ☐ Relatives of | □ Letter | ☐ Phone | □ Other | |
| | participants | | | (specify): | |
| | ☐ Others (please | □ Letter | ☐ Phone | □ Other | |
| | specify): | | | (specify): | |
| 4.5.02 | Please explain why contact | t is being m | ı<br>nade – appe | end copies of | relevant |
| | correspondence as suppor | rting eviden | ce | | |
| | If applicable | | | | |
| | - | | | | |
| 4.6 | Community Health Index | (CHI) Datab | oase Please | read section | 4.6 of the guidance |
| Comple | ete this section if access to C | HI Databas | e is required | d Not app | licable |
| 4.6.01 | What monitoring and audit of | of the use o | f | | |
| | CHI is planned? Please pro | vide details | | | |
| 4.6.02 | What technical method will | be used to | | | |
| | access CHI (online read-on | ly, downloa | d, | | |
| | other extract, anonymised e | extract, etc) | ? | | |
| | Please provide details | | | | |





| 4.6.03 Have any risks been identified in the |
|----------------------------------------------|
| proposal which relate specifically to |
| CHI? |



5.2.03

documentation



## Section 5 - Methodology & Data Processing

| | <u> </u> | |
|---|---|---|
| 5.1 | Methodology Please read section 5.1 of the guidance | |
| 5.1.01 | Does the proposal require any of the following: | |
| | oximes Data $oximes$ Single anonymised data extra | ct |
| | matching/linking | |
| | ☐ Use of matched | |
| | controls | |
| | Other (please specify): | |
| 5.1.02 | Who is carrying out any indexing/ | Data controler - national |
| | linkage/anonymisation, and where? | Services Scotland (@Farr |
| | | Institute) |
| 5.1.03 | Which data sources listed at section 4.1 and 4.2 will | Scottish Morbidity Record |
| | NSS/NRS receive identifiers for linkage purposes? | (SMR 01) |
| 5.1.04 | What variables will be provided for linkage? | |
| | X CHI Number Forename | □ Surname |
| | □ Date of Birth □ Address or Postcode | □ NHS Number |
| | Other Please Specify: | |
| 5.2 | Access Please read section 5.2 of the guidance | |
| Comple | te the following section if you answered 'No' to question 3.6. | 1 |
| 5.2.01 | At what location is identifiable or potentially identifiable | |
| | data being accessed? | |
| 5.2.02 | Please provide details of security policy/procedure | |
| | governing access to this physical and technical | |
| | environment – append supporting documentation | |

Does this policy/procedure cover password policy in

detail? Please provide details/ append supporting





| 5.2.04 | Does this policy/procedure cover user account | |
|---|---|---|
| | management, including review or removal of access to | |
| | sensitive/personal data, in detail? Please provide details/ | |
| | append supporting documentation | |
| 5.2.05 | Will individuals with access to data have individual or | |
| | shared accounts? | |
| 5.2.06 | Will the data be accessed by staff working off site eg staff | Choose an item. |
| | working from home at any time during the duration of the | |
| | proposal? | |
| 5.2.06b | If yes, are policies/procedures in place to facilitate, | If applicable |
| | monitor and audit this access? Please provide details/ | |
| | append supporting documentation | |
| 5.2.07 | Provide any additional detail of how data is protected | If applicable |
| | from unauthorised access | |

| 5.3 | Store & Use Please read section 5.3 of the guidance | |
|---|---|---|
| Comple | Complete the following section if you answered 'No' to question 3.6.1 | |
| 5.3.01 | Where is data being stored and used? (location, | |
| | organisation, address – refer to addresses in previous | |
| | sections if appropriate) | |
| 5.3.02 | Data Protection Registration Number | If applicable |
| 5.3.03 | ISO 27001 Cert. No. | If applicable |
| 5.3.04 | Please provide details of security policy/procedure | |
| | governing storage and use of data within this physical and | |
| | technical environment – append supporting | |
| | documentation | |
| 5.3.05 | Does this policy/procedure cover the implementation of | |
| | up-to-date controls for the detection and prevention of | |
| | malware? Please provide details/ append supporting | |
| | documentation | |
| 5.3.06 | Does this policy/procedure cover access control and | |
| | auditing of system administrator activity? Please provide | |
| | details/ append supporting documentation | |





| 5.3.07 | Does this policy/procedure cover the production of |
|---|---|
| | backups and the controls in place around these? Please |
| | provide details/ append supporting documentation |
| 5.3.08 | Does this policy/procedure describe the controls in place |
| | to prohibit unauthorised copying of data? Please provide |
| | details/ append supporting documentation |
| 5.3.09 | Does this policy/procedure describe physical and site |
| | controls? Please provide details/ append supporting |
| | documentation |
| 5.3.10 | Does this policy/procedure cover hardware repair, |
| | replacement or disposal and protection of data from |
| | inappropriate access during such procedures? Please |
| | provide details/ append supporting documentation |
| 5.3.11 | Describe the systems, software and security used to store |
| | and use data - please provide details/ append supporting |
| | documentation |
| 5.3.12 | Is outsourced IT in use? Please give details |
| Please | repeat section 5.3 above for each relevant location in the proposal – see guidance |

| 5.4 | Transfer Please read section 5.4 of the guidance | |
|---|---|---|
| 5.4.01 | Please provide details of security policy/procedure to | Identifiable data will not be |
| | ensure that data will be transferred in such a way that it is | transported. Only results |
| | protected from inappropriate or unauthorised access | from statistical analyses will |
| | (mention email encryption, secure file transfer protocols | be downloaded through |
| | SFTP, device encryption, physical controls, etc, as | secure file transfer |
| | appropriate) - append supporting documentation | protocols while connecting |
| | | to the safe haven. |
| | | Downloaded data will be |
| | | stored solely on computer |
| | | at the Radboud University |
| | | Medical Center, complying |





| | | to its electronic safety |
|---|---|---|
| | | protocols. |
| 5.4.02 | At what intervals/ trigger points will data transfer take | Analysed data will be |
| | place? | transferred regularly, during |
| | | a period of 4 months. |
| 5.4.03 | Will any identifiable or potentially identifiable data be | No |
| | transferred outside of the UK? | |
| 5.4.03b | If yes, please provide details of the country of destination, | If applicable |
| | the method of transfer, the proposed location and method | |
| | of storage outside of the UK, and details of any further | |
| | onward transfer | |
| 5.4.04 | Other than initial transfers from source systems, is there | No |
| | any copying of data required within the proposal? Please | |
| | give details | |
| 1 | | I I |

| 5.5 | Dissemination Please read section 5.5 of the guidance | |
|---|---|---|
| 5.5.01 | Will proposal findings be published or disseminated | Yes |
| | beyond the proposal team? | |
| 5.5.01a | If yes, how will proposal findings be published or | Results will be published |
| | disseminated, to what audience and in what format? | as a paper in a peer- |
| | Please give details | reviewed medical journal. |
| | | Results will further be |
| | | presented a surgical |
| | | conferences and |
| | | congresses using |
| | | powerpoint format. |
| 5.5.01b | If yes, what steps will be taken to ensure that persons | Graphs and tables in |
| | cannot be identified in published findings (eg disclosure | publications will provide |
| | control procedures (safe haven), use of aliases, | only large nationwide |
| | numbers, avoidance of small geographical areas, | number that is not |
| | avoidance of small numbers , etc)? Please give details | identifiable. |
| 5.5.01c | If yes, are there any circumstances where a living or | No |
| | dead individual would be cited? (eg where a person | |





| | consented to their data being used as a case study)? | |
|---------|----------------------------------------------------------|----|
| | Please give details | |
| 5.5.01d | If yes, were any permissions to publish data required or | No |
| | sought (for example from data controllers)? Please | |
| | provide details | |

| 5.6 | Retain/Dispose Please read section 5.6 of the guidance |
|--------|--------------------------------------------------------------|
| 5.6.01 | Which information/data/records retention policy will you be |
| | applying to the proposal data (details of the policy and the |
| | organisation to which it belongs)? |
| 5.6.02 | How long do you intend to retain identifiable or potentially |
| | identifiable data after the conclusion of the proposal |
| | (including archive/backup copies)? |
| 5.6.03 | Who will retain the data and where? |
| 5.6.04 | What is the purpose for retaining the data for the specified |
| | time? |
| 5.6.05 | What method of disposal or destruction will be used when |
| | this period has expired (including archive/backup copies)? |
| 5.6.06 | What evidence will be obtained that destruction has |
| | occurred (eg IT supplier certificate of destruction, etc)? |

| 5.7 | Review Please read section 5.7 of the guidance |
|---|---|
| 5.7.01 | Describe how the mechanisms which safeguard data |
| | security will be audited and reviewed at regular intervals to |
| | ensure their continued efficacy |
| 5.7.02 | Describe any resource implications to any of the proposed |
| | measures for the protection of physical or technical |
| | security of information which are unresolved at the time of |
| | this application? (for example encryption of devices is an |
| | intention not yet fulfilled, training is not yet undertaken, etc) |
| 5.7.03 | Describe the breach reporting mechanisms to be invoked |
| | in the event of any inappropriate access to data or other |
| | information security incident |









#### Section 6 - Declaration

- I DECLARE THAT this application is accurate, and that, should it be successful, any health
  data made accessible will be used for no other purpose, and in no other way, than as
  described above.
- I UNDERTAKE TO notify the Public Benefit and Privacy Panel of any future changes to the purpose or manner in which data is processed in accordance with this application.
- I UNDERSTAND THAT any future applications by me, or my employing or sponsoring organisation, may be refused should any health data made accessible be used for any other purpose or in any other way than that described above.
- I CERTIFY THAT all those who have access to health data in this proposal are aware of
  the requirements of confidentiality and understand that any breach (eg disclosure of
  confidential information to a person not authorised to receive it) will be reported to the data
  controller, and in the case of NHS Scotland originated data to Scottish Government
  eHealth division.
- I GUARANTEE THAT no publication will appear in any form in which an individual may be identified without the written permission of that individual, and that I will apply appropriate disclosure control when planning publications involving the data requested.
- I UNDERSTAND THAT the Data Controller, and agents acting on its behalf, reserves the right to inspect the data on the sites where it is being processed.

To be signified by the APPLICANT

Name (in Capitals): RICHARD TEN BROEK Date: 22-04-2018

I DECLARE THAT (the applicant named above) is a bona fide worker engaged in a
reputable project and that the data he/she asks for can be entrusted to him/her in the
knowledge that he/she will conscientiously discharge his/her obligations, including in
regard to confidentiality of the data, as stated in the declaration above.

To be signified by the INFORMATION CUSTODIAN named in Section 1.3 above (where the Information Custodian is not the applicant).

Lon Block





| Name (in Capitals): | Date: |
|---------------------|-------|

## Section 7 - Supporting Evidence

## Supporting Evidence Please read section 7 of the guidance

Please list each piece of supporting evidence which you have included with your application in the box below – the name of each should clearly indicate what the document/file/reference is about

- Appendix with list of OPCS 4.7 and ICD10 codes relevant for selection of data
- Certificates of Research data and confidentiality training
- Protocol as send for IRB approval
- IRB approval
- Privacy Impact assessment





## Appendix A - Reference lists for applicants

| 1. Examples of Existing Datasets and Data Sources | |
|---|---|
| SMR 00 Outpatients | SMR 04 Mental Health |
| SMR 01 Inpatients and Day Cases | SMR 06 Cancer Registration |
| SMR 02 Maternity | SMR 11/SBR Neonatal/Scottish Birth |
| | Records |
| Scottish Drugs Misuse Database (SDMD) | Birth Registrations |
| A&E – Accident & Emergency | Stillbirth Registrations |
| PIS Prescribing Information | Death Registrations |
| CHSP-PS/CHSP-S/SIRS – Child Health | <u>SCI-DC</u> |
| Surveillance and Immunisation | |

NHS National Service Scotland's Information Services Division (ISD) maintains a <u>National</u> <u>Dataset Catalogue (NDC)</u> containing details of all health and health related datasets that are held by ISD. The Administrative Data Liaison Service (ADLS) publishes further information on key <u>NHSScotland datasets</u>

| 2. Common Identifiable Variables | | |
|---|---|---|
| Forename | Middle Name | Surname |
| CHI Number | Date of Birth | UK NHS Birth Registration Number |
| Gender | Postcode | |

| 3. Recognised Safe Havens |
|---------------------------------------------------------------------------|
| NHS NSS ISD Electronic Data Research Innovation Service (@Farr Institute) |
| NHS Research Scotland South East (ACCORD) |
| NHS Research Scotland East (TASC) |
| NHS Research Scotland North (DaSH) |
| NHS Research Scotland West |
| University of Dundee Health Informatics Centre (HIC) |
| National Records Scotland Scottish Longitudinal Study (SLS) |
| Robertson Centre @ Glasgow University |





## 4. Research and Information Governance Training

MRC Research Data and Confidentiality online module

University of Edinburgh SHIP Information Governance training

NHS Health and Social Care Information Centre On-line Information Governance training

NHSScotland Information Governance eLearning:

- Safe Information Handling (Foundation Level)
- Information Handling in Practice (Intermediate Level)

| 5. Sensitive Data Categories | | |
|---|---|---|
| Abortion | Mental health | Contraception |
| Pregnancy in age < 16 years | Drugs and alcohol misuse | Crime related statistics |
| Sexually transmitted disease | Suicide | Ethnicity |
| Assisted conception | | |

| 6. Vulnerable Populations | |
|---------------------------|--------------------------------|
| Adults with Incapacity | Drugs users |
| Minority ethnic groups | Specific religious affiliation |





## Appendix B –The Caldicott Principles & the Data Protection Principles (& Schedules)

## 1. Caldicott Principles

### 1. Justify the purpose(s)

Every single proposed use or transfer of patient identifiable information within or from an organization should be clearly defined and scrutinized, with continuing uses regularly reviewed, by an appropriate guardian.

## 2. Don't use patient identifiable information unless it is necessary

Patient identifiable information items should not be included unless it is essential for the specified purpose(s) of that flow. The need for patients to be identified should be considered at each stage of satisfying the purpose(s).

## 3. Use the minimum necessary patient-identifiable information

Where use of patient identifiable information is considered to be essential, the inclusion of each individual item of information should be considered and justified so that the minimum amount of identifiable information is transferred or accessible as is necessary for a given function to be carried out.

4. Access to patient identifiable information should be on a strict need-to-know basis
Only those individuals who need access to patient identifiable information should have
access to it, and they should only have access to the information items that they need to see.
This may mean introducing access controls or splitting information flows where one
information flow is used for several purposes.

# 5. Everyone with access to patient identifiable information should be aware of their responsibilities

Action should be taken to ensure that those handling patient identifiable information - both clinical and non-clinical staff - are made fully aware of their responsibilities and obligations to respect patient confidentiality.

## 6. Understand and comply with the law

Every use of patient identifiable information must be lawful. Someone in each organization





handling patient information should be responsible for ensuring that the organization complies with legal requirements.

# 7. The duty to share information can be as important as the duty to protect patient confidentiality

Health and social care professionals should have the confidence to share information in the best interests of their patients within the framework set out by these principles. They should be supported by the policies of their employers, regulators and professional bodies.

### 2. Data Protection Principles

- Personal data shall be processed fairly and lawfully and, in particular, shall not be processed unless –
  - (a) at least one of the conditions in Schedule 2 is met, and
  - (b) in the case of sensitive personal data, at least one of the conditions in Schedule 3 is also met
- 2. Personal data shall be obtained only for one or more specified and lawful purposes, and shall not be further processed in any manner incompatible with that purpose or those purposes
- **3.** Personal data shall be adequate, relevant and not excessive in relation to the purpose or purposes for which they are processed
- 4. Personal data shall be accurate and, where necessary, kept up to date
- **5.** Personal data processed for any purpose or purposes shall not be kept for longer than is necessary for that purpose or those purposes
- **6.** Personal data shall be processed in accordance with the rights of data subjects under this Act
- 7. Appropriate technical and organizational measures shall be taken against unauthorized or unlawful processing of personal data and against accidental loss or destruction of, or damage to, personal data





8. Personal data shall not be transferred to a country or territory outside the European Economic Area unless that country or territory ensures an adequate level of protection for the rights and freedoms of data subjects in relation to the processing of personal data

#### 3. Data Protection Schedule 2 & 3 Conditions

### Schedule 2 - Conditions for Processing any Personal Data

- 1. The data subject has given his **consent** to the processing
- 2. The processing is necessary—
  - (a) for the **performance of a contract** to which the data subject is a party, or
  - (b) for the taking of steps at the request of the data subject with a view to entering into a contract
- 3. The processing is necessary for compliance with any **legal obligation** to which the data controller is subject, other than an obligation imposed by contract
- 4. The processing is necessary in order to protect the vital interests of the data subject
- 5. The processing is necessary—
  - (a) for the administration of justice,
  - (aa) for the exercise of any functions of either **House of Parliament**,
  - (b) for the exercise of any functions conferred on any person by or under any **enactment**,
  - (c) for the exercise of any functions of the Crown, a Minister of the Crown or a government department, or
  - (d) for the exercise of any other functions of a **public nature exercised in the public interest** by any person
- 6. (1) The processing is necessary for the purposes of **legitimate interests** pursued by the data controller or by the third party or parties to whom the data are disclosed, except where the processing is unwarranted in any particular case by reason of prejudice to the rights and freedoms or legitimate interests of the data subject.
- (2) The Secretary of State may by order specify particular circumstances in which this condition is, or is not, to be taken to be satisfied

#### Schedule 3 – Conditions for Processing any Sensitive Personal Data

1. The data subject has given his explicit consent to the processing of the personal data





- 2. (1) The processing is necessary for the purposes of exercising or performing any right or obligation which is conferred or imposed by law on the data controller in connection with **employment**
- 3. The processing is necessary—
  - (a) in order to protect the **vital interests** of the data subject or another person, in a case where—
    - (i) consent cannot be given by or on behalf of the data subject, or
    - (ii) the data controller **cannot reasonably be expected to obtain the consent** of the data subject, or
  - (b) in order to protect the **vital interests** of another person, in a case where **consent** by or on behalf of the data subject has been **unreasonably withheld**
- 4. The processing—
  - (a) is carried out in the course of its legitimate activities by any body or association which—
    - (i) is not established or conducted for profit, and
    - (ii) exists for political, philosophical, religious or trade-union purposes,
  - (b) is carried out with appropriate safeguards for the rights and freedoms of data subjects,
  - (c) relates only to individuals who either are members of the body or association or have regular contact with it in connection with its purposes, and
  - (d) does not involve disclosure of the personal data to a third party without the consent of the data subject
- 5. The information contained in the personal data has been **made public** as a result of steps deliberately taken **by the data subject**
- 6. The processing—
  - (a) is necessary for the purpose of, or in connection with, any **legal proceedings** (including prospective legal proceedings),
  - (b) is necessary for the purpose of obtaining legal advice, or
  - (c) is otherwise necessary for the purposes of establishing, exercising or defending **legal rights**
- 7. (1) The processing is necessary—
  - (a) for the administration of justice,
  - (aa) for the exercise of any functions of either House of Parliament,
  - (b) for the exercise of any functions conferred on any person by or under an **enactment**, or





- (c) for the exercise of any functions of the Crown, a Minister of the Crown or a government department
- (2)The Secretary of State may by order—
  - (a) exclude the application of sub-paragraph (1) in such cases as may be specified, or
  - (b) provide that, in such cases as may be specified, the condition in sub-paragraph (1) is not to be regarded as satisfied unless such further conditions as may be specified in the order are also satisfied

## 7A. (1) The processing—

- (a) is either—
  - (i) the disclosure of sensitive personal data by a person as a member of an **anti-fraud** organisation or otherwise in accordance with any arrangements made by such an organisation; or
  - (ii) any other processing by that person or another person of sensitive personal data so disclosed; and
- (b) is necessary for the purposes of preventing fraud or a particular kind of fraud
- (2) In this paragraph "an anti-fraud organisation" means any unincorporated association, body corporate or other person which enables or facilitates any sharing of information to prevent fraud or a particular kind of fraud or which has any of these functions as its purpose or one of its purposes
- 8. (1) The processing is necessary for **medical purposes** and is undertaken by—
  - (a) a health professional, or
  - (b) a person who in the circumstances owes a duty of confidentiality which is equivalent to that which would arise if that person were a health professional
- (2) In this paragraph "medical purposes" includes the purposes of preventative medicine, medical diagnosis, medical research, the provision of care and treatment and the management of healthcare services
- 9. (1) The processing—
  - (a) is of sensitive personal data consisting of information as to racial or ethnic origin,
  - (b) is necessary for the purpose of identifying or keeping under review the existence or absence of **equality of opportunity** or treatment between persons of different racial or ethnic origins, with a view to enabling such equality to be promoted or maintained, and
  - (c) is carried out with appropriate safeguards for the rights and freedoms of data subjects





- (2) The Secretary of State may by order specify circumstances in which processing falling within sub-paragraph (1)(a) and (b) is, or is not, to be taken for the purposes of sub-paragraph (1)(c) to be carried out with appropriate safeguards for the rights and freedoms of data subjects
- 10. The personal data are processed in circumstances specified in an order made by the Secretary of State for the purposes of this paragraph